CLINICAL TRIAL: NCT02650843
Title: Non-motor Symptoms and Brain Dopamine Transporter Binding: An Observational Study in Parkinsonism
Brief Title: Non-motor Symptoms and Brain Dopamine Transporter Binding
Acronym: NMDAT
Status: Active, not recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: T12/2014
Record Dates: First submitted 2016-01-05; First posted 2016-01-08 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease; Parkinsonism
Keywords: Parkinsonism; DAT Dopamine transporter; SPECT
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with parkinsonism: Patients with parkinsonism that are referred for DAT SPECT imaging in Turku University Hospital, Finland or Helsinki University Hospital, Finland
  Interventions: Other: DAT SPECT imaging

INTERVENTIONS:
Other: DAT SPECT imaging

SUMMARY:
This project aims to clarify the role non-motor symptoms in the development of Parkinson's disease (PD) and to improve diagnostics at very early stages of PD. The project involves multidimensional measures of disease biomarkers together with brain dopamine transporter (DAT) imaging with [123I]FP-CIT single photon emission computed tomography (SPECT).

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Age 18-100 years
* Referred for clinical DAT SPECT in Turku or Helsinki

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with parkinsonism
Sampling Method: Non-Probability Sample
Enrollment: 455 (Actual)
Dates: Start 2015-01; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
DAT SPECT striatal specific binding ratio | Up to 10 years

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Eklund M, Nuuttila S, Joutsa J, Jaakkola E, Makinen E, Honkanen EA, Lindholm K, Vahlberg T, Noponen T, Ihalainen T, Murtomaki K, Nojonen T, Levo R, Mertsalmi T, Scheperjans F, Kaasinen V. Diagnostic value of micrographia in Parkinson's disease: a study with [123I]FP-CIT SPECT. J Neural Transm (Vienna). 2022 Jul;129(7):895-904. doi: 10.1007/s00702-022-02517-1. Epub 2022 May 27. PMID 35624405
- [Derived] Nuuttila S, Eklund M, Joutsa J, Jaakkola E, Makinen E, Honkanen EA, Lindholm K, Noponen T, Ihalainen T, Murtomaki K, Nojonen T, Levo R, Mertsalmi T, Scheperjans F, Kaasinen V. Diagnostic accuracy of glabellar tap sign for Parkinson's disease. J Neural Transm (Vienna). 2021 Nov;128(11):1655-1661. doi: 10.1007/s00702-021-02391-3. Epub 2021 Jul 30. PMID 34328563